CLINICAL TRIAL: NCT05798715
Title: Comparative, Randomized, Single Dose, Two-way Crossover Bioequivalence Study to Determine the Bioequivalence of Metformin HCl From Gleptomet 50/1000 mg F.C.Tablets (EVA Pharma for Pharmaceuticals & Medical Appliances, Egypt) and Janumet 50/1000 mg F.C.Tablets (Merck Sharp & Dohme, The Netherlands) After a Single Oral Dose Administration of Each to Healthy Adults Under Fed Conditions.
Brief Title: Bioequivalence Study of of Metformin HCl From Gleptomet 50/1000 mg F.C.Tablets (EVA Pharma, Egypt) and Janumet 50/1000 mg F.C.Tablets (Merck Sharp & Dohme, The Netherlands)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genuine Research Center, Egypt (Industry)
Collaborators: Eva Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: GRC/1/21/1044
Record Dates: First submitted 2023-03-22; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Healthy
MeSH Terms: interventions — Sitagliptin Phosphate; Sitagliptin Phosphate, Metformin Hydrochloride Drug Combination

STUDY DESIGN:
Intervention Model Description: Comparative, Randomized, Single Dose, Two-way Crossover Bioequivalence Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T test (Experimental): 1 tablet contains 1000 mg Metformin HCl & 50 mg Sitagliptin orally administrated with 240 mL of a 20% glucose solution in water, followed by 60 mL of the glucose solution administered every 15 min for up to 4 hours after dosing
  Interventions: Drug: Gleptomet 50/1000(Metformin HCl & Sitagliptin)
- R Reference (Active Comparator): 1 tablet contains 1000 mg Metformin HCl & 50 mg Sitagliptin orally administrated with 240 mL of a 20% glucose solution in water, followed by 60 mL of the glucose solution administered every 15 min for up to 4 hours after dosing
  Interventions: Drug: Janumet 50/1000(Metformin HCl & Sitagliptin)

INTERVENTIONS:
Drug: Gleptomet 50/1000(Metformin HCl & Sitagliptin) — Test drug
  Other Names: Janumet
  Arms: T test
Drug: Janumet 50/1000(Metformin HCl & Sitagliptin) — Reference drug
  Other Names: Janumet
  Arms: R Reference

SUMMARY:
Comparative, Randomized, Single Dose, Two-way Crossover Bioequivalence Study to determine the bioequivalence of Metformin HCl From Gleptomet 50/1000 mg F.C.Tablets (EVA Pharma, Egypt) and Janumet 50/1000 mg F.C.Tablets (Merck Sharp & Dohme, The Netherlands)

DETAILED DESCRIPTION:
Healthy volunteers, 18-55 years of age, selected from the Egyptian population fulfilling the selection criteria. All dosed subject samples will be analyzed and their data will be included in the final study report.

Primary Pharmacokinetic Parameters: Cmax, AUC0→t and AUC0→∞ Secondary Pharmacokinetic Parameters: Ke, tmax and t1/2e. ANOVA using 5% significance level for transformed (with the 90% confidence intervals) and untransformed data of Cmax, AUC0→t and AUC0→∞ and for untransformed data of Ke, tmax and t1/2e.

The confidence intervals of logarithmically transformed Test/Reference ratios for Cmax, AUC0→t and AUC0→∞ to be within 80.00-125.00%.

A comprehensive final report will be issued upon the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female, age 18 to 55 years, inclusive.
2. Body weight within 15% of normal range (18.5-30.0) according to the accepted normal values for body mass index (BMI).
3. Medical demographics without evidence of clinically significant deviation from normal medical condition, eg.: no history of heart, liver, kidney, gastrointestinal, nervous system, or metabolic abnormalities.
4. Results of clinical laboratory test are within the normal range or with a deviation that is not considered clinically significant by principal investigator.
5. Females should be on a suitable birth control method.
6. Fully informed subjects that consented to participate in the study.

Exclusion Criteria:

1. Subjects with known allergy to the products tested.
2. Subjects who meet any of the contraindications to the administration of Sitagliptin and/or Metformin HCl.
3. Subjects who are going to get an injection of dye or contrast agents for an x-ray procedure.
4. Subject does not agree not to consume any medication or food which may affect CYP3A4 enzyme at least one week prior to first study drug administration until donating the last sample of the study.
5. Subjects that do not agree not to consume alcohol-containing beverages and foods for 1 week before dosing and throughout the period of sample collection.
6. Heavy smokers.
7. Female subjects who were pregnant or nursing.
8. Acute infection within one week preceding first study drug administration.
9. History of drug or alcohol abuse.
10. Subject does not comply with the stated instruction of not taking any prescription or non-prescription drugs within two weeks before first study drug administration and until the end of the study.
11. Subject is on a special diet (for example subject is vegetarian).
12. Subject does not agree not to consume any beverages or foods containing methyl-xanthenes e.g. caffeine (coffee, tea, cola, chocolate etc.) 48 hours prior to the study administration of either study period until donating the last sample in each respective period.
13. Subject does not agree not to consume any beverages or foods containing grapefruit 7 days prior to first study drug administration until the end of the study.
14. Subject has a family history of severe diseases which have direct impact on the study.
15. Participation in a bioequivalence study or in a clinical study within the last 60 days, before first study drug administration.
16. Subject intends to be hospitalized within 3 months after first study drug administration.
17. Subjects who have blood donated or lost more than 500 mL blood within 3 months prior to the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Cmax | Up to 36 hours post dose in each treatment period
  to measure the maximal measured plasma concentration

SECONDARY OUTCOMES:
Tmax | Up to 36 hours post dose in each treatment period
  time of the maximum plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elshafeey, Ph.D. Pharma, Study Director — Genuine Research Center
Locations (1):
- Genuine Research Center GRC, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chow SC, Wang H. On sample size calculation in bioequivalence trials. J Pharmacokinet Pharmacodyn. 2001 Apr;28(2):155-69. doi: 10.1023/a:1011503032353. PMID 11381568
- [Background] Schuirmann DJ. A comparison of the two one-sided tests procedure and the power approach for assessing the equivalence of average bioavailability. J Pharmacokinet Biopharm. 1987 Dec;15(6):657-80. doi: 10.1007/BF01068419. PMID 3450848
- [Background] Diletti E, Hauschke D, Steinijans VW. Sample size determination for bioequivalence assessment by means of confidence intervals. Int J Clin Pharmacol Ther Toxicol. 1991 Jan;29(1):1-8. PMID 2004861